CLINICAL TRIAL: NCT06522347
Title: Mycobacteria Registry Study: Prospective Observational Study in Austria
Status: Recruiting | Type: Observational
Sponsor: Ludwig Boltzmann Institute for Lung Health (Other)
Collaborators: Sigmund Freud PrivatUniversitat (Other)
Responsible Party: Principal Investigator, Robab Breyer-Kohansal, Prim.a Priv.-Doz.in Dr.in, Ludwig Boltzmann Institute for Lung Health
Other Study IDs: TBC-NTM
Record Dates: First submitted 2024-07-22; First posted 2024-07-26 (Actual); Last update posted 2024-07-26 (Actual); Status verified 2024-07

CONDITIONS: Non-Tuberculous Mycobacterial Pneumonia; Tuberculosis
Keywords: Mycobacterium tuberculosis; Nontuberculous Mycobacteria; Mycobacterium Infections
MeSH Terms: conditions — Tuberculosis; Mycobacterium Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this non-interventional registry study is to systematically collect epidemiological and clinical data throughout the treatment course to learn about effectiveness of treatments. We will document the natural course of therapy without additional interventions. The main question to answer is:

What are the risk factors for mortality due to infection with Mycobacteria tuberculosis (TB) or Nontuberculous mycobacteria (NTM) in Austria?

Data from participants already receiving treatment as part of their regular medical care for TB or NTM infections will be collected.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with Mycobacterium tuberculosis or non-tuberculous mycobacteria infection
* individuals aged 18 years or older
* written informed consent

Exclusion Criteria:

* to not comprehend and rightfully judge participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient presenting to outpatient clinic or ward of Klink Penzing or Klinik Hietzing due to Mycobacteria infection.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2053-12-31 (Estimated); Study Completion 2053-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 years
  Mortality due to tuberculosis or NTM infection in Austria

SECONDARY OUTCOMES:
Prevalence | 30 years
  Prevalence of mycobacterial infections in Austria
Patient cohort | 30 years
  Description of the patient cohort
Risk factors | 30 years
  Identification of risk factors for treatment failure and complications

CONTACTS AND LOCATIONS:
Locations (3):
- Austria (3):
  - Klinik Hietzing, Vienna
  - Klinik Penzing, Vienna
  - Ludwig Boltzmann Institut for Lung Health, Vienna